CLINICAL TRIAL: NCT05817019
Title: A Double-blind, Randomized, Parallel Design Study to Compare Postoperative Recovery Between the Sugammadex Group and the Neostigmine Group in Patients After COVID-19.
Brief Title: Postoperative Sugammadex After COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Min, Too Jae, Professor, Korea University Ansan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023AS0079
Record Dates: First submitted 2023-04-11; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: General Anesthesia; COVID-19
Keywords: COVID-19; Postoperative Complications
MeSH Terms: conditions — COVID-19; Postoperative Complications | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, parallel design study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The neuromuscular reversal agent is received and prepared in advance by a separate medical staff (a separate anesthesiologist who does not participate in the patient's anesthesia), and the corresponding prescription order is made separately when the patient leaves the recovery room. Since it is diluted with physiological saline and prepared in a total amount of 5cc, the patient and the patient's anesthetist do not know about the drug until they leave the recovery room (double-blinded).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Experimental): sugammadex 2mg/kg
  Interventions: Drug: Sugammadex Sodium
- Neostigmine (Active Comparator): neostigmine 50µg/kg + glycopyrollate 0.01mg/kg
  Interventions: Drug: neostigmine 50µg/kg + glycopyrollate 0.01mg/kg

INTERVENTIONS:
Drug: Sugammadex Sodium — Sugammadex Sodium 2mg/kg when TOF >= 2, postoperative period
  Other Names: Bridion
  Arms: Sugammadex
Drug: neostigmine 50µg/kg + glycopyrollate 0.01mg/kg — neostigmine 50µg/kg + glycopyrollate 0.01mg/kg when TOF >= 2, postoperative period
  Other Names: neostigmine
  Arms: Neostigmine

SUMMARY:
Researcher want to compare and evaluate the effect of sugammadex on postoperative recovery, with a focus on the occurrence of postoperative urinary dysfunction, in patients who have undergone regular abdominal surgery within a year of being infected with and treated for COVID-19.

Post COVID-19 condition is a new and poorly understood clinical syndrome with potentially significant and life-altering consequences. Recent studies suggest that patients who have recovered from COVID-19 may experience autonomic dysfunction and be at risk for autonomic dysregulation/syndrome. In most patients undergoing general anesthesia, neuromuscular blockers are used, and their residual effects delay the recovery of autonomic function after surgery, leading to problems such as worsening bladder and bowel function. Therefore, reversal agents are used to aid in postoperative muscle recovery, with sugammadex and neostigmine being commonly used in clinical practice. While sugammadex is generally expected to result in faster postoperative recovery, limited reports exist on its effectiveness in patients who have recovered from COVID-19. This study aims to verify whether sugammadex is more effective than neostigmine in aiding the recovery of bowel and pulmonary function after surgery in patients who have recovered from COVID-19.

DETAILED DESCRIPTION:
The COVID-19 has had a huge impact on the world, infected tens of millions and killed hundreds of thousands, and has become a threat to humanity's medical defense system. COVID-19 was understood as an acute infection among infections, and it was expected that there would be little or no other risk if the acute symptoms were treated. Contrary to our expectations, however, patients with a history of infection with the coronavirus have reported patients with sequelae lasting for more than several months. The symptoms shown by these patients were not limited to some tissues and organs, but were distributed in various ways throughout our body. These symptoms were defined as 'long COVID'. In particular, among the symptoms of long COVID patients, there were patients who were diagnosed with orthostatic hypotension, vasovagal syncope, and orthostatic tachycardia syndrome from symptoms such as palpitations, shortness of breath, and chest pain. What these diseases have in common is that they are autonomic nervous system diseases. Therefore, it can be assumed that long COVID patients have damage to the function of the autonomic nervous system due to past infections, and many studies have been conducted on this.

The main components of general anesthesia are known to be unconsciousness, muscle relaxation, analgesia, and reflex suppression. Among these, the reasons why muscle relaxation is necessary in general anesthesia include ease of intubation and suppression of unnecessary patient movements during surgery to create a suitable environment for surgery. For muscle relaxation, anesthesiologists administer neuromuscular relaxants, mainly non-depolarizing muscle relaxants. Neuromuscular relaxants have the role of inhibiting neurotransmission by acting on the motor nerve endings of skeletal muscles, because they act on nicotinic cholinergic receptors in motor nerve endings. However, neuromuscular relaxants also act on muscarinic cholinergic receptors to inhibit neurotransmission. Since these muscarinic cholinergic receptors are distributed in the parasympathetic nerves of the autonomic nervous system, neuromuscular relaxants also inhibit the autonomic nerve system controlled by the parasympathetic nerves.

Since neuromuscular relaxants are eliminated from the body by pharmacokinetics, the function of the autonomic nervous system, which has been suppressed by using neuromuscular relaxants, gradually recovers over time. However, if the action of a neuromuscular relaxant remains after surgery, the patient will experience autonomic dysfunction even after surgery, which causes considerable discomfort to the patient. Among them, the symptoms of autonomic dysfunction related to the parasympathetic nerve that patients mainly feel are related to the bladder and bowel. Therefore, after the surgery, the anesthesiologist performs the process of reversing the action of the neuromuscular relaxant when ending general anesthesia, which makes it possible to expect the recovery of the patient's autonomic nervous system function.

There are two main mechanisms of the drugs used for reversal of nondepolarizing neuromuscular relaxants. First, there is a drug that inhibits the action of the neuromuscular relaxant by directly attaching to the neuromuscular relaxant, and second, there is a drug that competitively inhibits the neuromuscular relaxant by increasing the amount of ach in the neuromuscular junction. In the meantime, many studies have shown that a drug with the former mechanism (sugammadex) is superior to the latter drug (typically neostigmine) in the recovery of patients after surgery. However, there is a lack of research on whether the same research results will be shown in long COVID patients who have caused damage to the autonomic nervous system.

Therefore, in this study, sugammadex and neostigmine as described above are divided and administered to approximately 300 long COVID patients in a double-blind manner, and the degree of urinary retention is compared to prove that sugammadex is superior to neostigmine in postoperative recovery even for long COVID patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 19 and 70 Male and Female All ethnicity Patients who are scheduled to take non-emergency abdominal surgery under general anesthesia.

Patients who had the diagnosis of covid-19 by PCR, hospitalized, and applied O2 supplement therapy.

ASA classification ≤ 3 Patients who had Covid-19 PCR positive within 1 year Patients who had hospitalized by Covid-19, followed by O2 therapy (nasal prong, continuous positive airway pressure (CPAP), ventilator etc.) Patients who hospitalized more than 48 hours after surgery. Patients who had a surgery for more than 1 hour.

Exclusion Criteria:

* Not meeting inclusion criteria Declined to participate Active Covid-19 patients with PCR positive. Patients are under 19 or over 70 years old

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
urinary retention incidence | postoperative 1 hour
  urinary retention incidence

SECONDARY OUTCOMES:
surgery time and anesthesia time | perioperative period
  surgery time and anesthesia time
recovery time after anesthesia | postoperative period, within 1 hour
  recovery time after anesthesia
intraoperative blood loss | perioperative period
  estimated blood loss
perioperative vital signs | perioperative period
  serial follow up during surgery and postoperative recovery room
additional sugammadex administration | postoperative period, within 1 hour
  incidence and dosage
bladder volume evaluated | postoperative 1 hour
  Sono-calculated (summation of self-voiding volume during self-voiding)
recovery score | postoperative 1 hour
  postoperative recovery score at PACU
pain score | postoperative 1 hour
  NRS
urinary retention | postoperative 24 and 48 hour
  presence of complication
acute lesion on chest X-ray | 2 days after surgery
  presence of complication
actual dosage of drugs for pain and nausea control | postoperative period, within 1 hour
  pain (ketorolac, fentanyl, tramadol, acetaminophen, nalbuphine, pethidcine, ketoprofen, propacetamol) nausea(ramosetron, metoclopramide, palonosetron)
other intraoperative events (awakening (eye opening), involuntary movement, occurrence of adverse events and unexpected side effects, etc.) | perioperative period
  presence of complication

CONTACTS AND LOCATIONS:
Overall Officials: Too Jae Min, M.D., Ph.D., Study Chair — Korea University Ansan Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT05817019/Prot_SAP_000.pdf